CLINICAL TRIAL: NCT01230385
Title: Randomized, Open-Label, Parallel Group Study To Investigate The Safety And Tolerability Of Multiple Dose Lersivirine (Proposed Phase 3 Formulation) For 21 Days In Healthy Subjects
Brief Title: Safety And Tolerability Of Multiple Dose Lersivirine For 21 Days In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5271049
Record Dates: First submitted 2010-10-08; First posted 2010-10-29 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Volunteers
Keywords: lersivirine; UK-453; 061; safety; tolerability; pharmacokinetics; HIV; non-nucleoside reverse transcriptase inhibitor; NNRTI
MeSH Terms: interventions — UK 453,061

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lersivirine 500 mg QD fasted (wet granulated tablet) (Experimental)
  Interventions: Drug: Lersivirine
- Lersivirine 500 mg QD fed (wet granulated tablet) (Experimental)
  Interventions: Drug: Lersivirine
- Lersivirine 750 mg QD fasted (wet granulated tablet) (Experimental)
  Interventions: Drug: Lersivirine
- Lersivirine 750 mg QD fed (wet granulated tablet) (Experimental)
  Interventions: Drug: Lersivirine
- Lersivirine 500 mg QD fasted (dry granulated tablet) (Active Comparator)
  Interventions: Drug: Lersivirine

INTERVENTIONS:
Drug: Lersivirine — Lersivirine 500 mg QD fasted (wet granulated tablet) for 21 days
  Arms: Lersivirine 500 mg QD fasted (wet granulated tablet)
Drug: Lersivirine — Lersivirine 500 mg QD fed (wet granulated tablet) for 21 days
  Arms: Lersivirine 500 mg QD fed (wet granulated tablet)
Drug: Lersivirine — Lersivirine 750 mg QD fasted (wet granulated tablet) for 21 days
  Arms: Lersivirine 750 mg QD fasted (wet granulated tablet)
Drug: Lersivirine — Lersivirine 750 mg QD fed (wet granulated tablet) for 21 days
  Arms: Lersivirine 750 mg QD fed (wet granulated tablet)
Drug: Lersivirine — Lersivirine 500 mg QD fasted (dry granulated tablet) for 21 days
  Arms: Lersivirine 500 mg QD fasted (dry granulated tablet)

SUMMARY:
Randomized, open-label, parallel group study in a group of 75 healthy subjects, to evaluate the safety and toleration of 2 different doses of lersivirine administered either fed or fasted (proposed Phase 3 formulation) given over 21 days, compared to lersivirine 500 mg QD (Phase 2b formulation). The pharmacokinetics of lersivirine in each group will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of multiple doses of lersivirine administered to healthy subjects over 21 days. | 21 days

SECONDARY OUTCOMES:
Lersivirine plasma pharmacokinetic parameter: AUC24, Cmax, C24, and Tmax on Day 7 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, New Haven, Connecticut, United States
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271049&StudyName=Safety%20And%20Tolerability%20Of%20Multiple%20Dose%20Lersivirine%20For%2021%20Days%20In%20Healthy%20Subjects%20